CLINICAL TRIAL: NCT02142595
Title: Comparison of the Postoperative Sleep Quality of Patients Sedation With i.v. Dexmedetomidine or Midazolam Undergoing Transurethral Prostatic Resection(TURP)
Brief Title: Postoperative Sleep Quality of Patients Sedation With i.v. Dexmedetomidine or Midazolam Undergoing TURP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, the Anesthesiology Department, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140515
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Quality of Patients Undergoing TURP
Keywords: dexmedetomidine; midazolam; sleep quality; delirium
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Delirium | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dexmeditomidine group D (Experimental): The sedative solution was prepared as a 10µg /ml dexmedetomidine in an unlabeled 20ml syringe. The sedative solution administered intravenously started at rate of kg (weight of patient)*0.6 ml/h over a 10-min period and then at rate of kg (weight of patient)*0.15 ml/h through syringe pump to the end of surgery
  Interventions: Drug: dexmedetomidine
- Midazolam group M (Experimental): The sedative solution was prepared as a 0.375mg/ml midazolam or normal saline in an unlabeled 20ml syringe. The sedative solution administered intravenously started at rate of kg (weight of patient)*0.6 ml/h over a 10-min period and then at rate of kg (weight of patient)*0.15 ml/h through syringe pump to the end of surgery
  Interventions: Drug: Midazolam
- group control (No Intervention): normal saline in an unlabeled 20ml syringe. The sedative solution administered intravenously started at rate of kg (weight of patient)*0.6 ml/h over a 10-min period and then at rate of kg (weight of patient)*0.15 ml/h through syringe pump to the end of surgery

INTERVENTIONS:
Drug: dexmedetomidine — The sedative solution administered intravenously started at rate of kg (weight of patient)*0.6 ml/h over a 10-min period and then at rate of kg (weight of patient)*0.15 ml/h through syringe pump to the end of surgery
  Arms: dexmeditomidine group D
Drug: Midazolam — The sedative solution administered intravenously started at rate of kg (weight of patient)*0.6 ml/h over a 10-min period and then at rate of kg (weight of patient)*0.15 ml/h through syringe pump to the end of surgery
  Arms: Midazolam group M

SUMMARY:
The investigators designed a study to determine whether dexmedetomidine versus midazolam combined with spinal anesthesia would provide same postoperative sleep quality in patients undergoing transurethral prostatic resection.

DETAILED DESCRIPTION:
The investigators designed a study to determine whether dexmedetomidine versus midazolam combined with spinal anesthesia would provide same postoperative sleep quality in patients undergoing transurethral prostatic resection.The bispectral index score (BIS) was monitored during the operation and the first postoperative night

ELIGIBILITY:
Inclusion Criteria:

* Participants were deemed eligible if they were candidates for spinal anesthesia undergoing TURP

Exclusion Criteria:

* The exclusion criteria were body mass index exceeding 30 kg/m2, preoperative Pittsburgh Sleep Quality Index global scores higher than 6, anesthesia time longer than 3 hours, allergy to drugs used in the study and treatment with sedatives and analgesics during the postoperative BIS-Vista monitoring period.

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Change of postoperative sleep quality | preoperation, first postoperative night
  The bispectral index score (BIS) was monitored during the operation and the first postoperative night

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,PhD., Study Director — Department of Anesthesiology the first hospital of CMU
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China